CLINICAL TRIAL: NCT01778803
Title: A Phase I/Ib Study of Paclitaxel in Combination With VS-6063, a Focal Adhesion Kinase Inhibitor, in Subjects With Advanced Ovarian Cancer
Brief Title: Phase I/Ib Study of Paclitaxel in Combination With VS-6063 in Patients With Advanced Ovarian Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Verastem, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VS-6063-101
Record Dates: First submitted 2013-01-22; First posted 2013-01-29 (Estimated); Last update posted 2017-05-17 (Actual); Status verified 2017-01

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — defactinib; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- defactinib (VS-6063) plus paclitaxel (Experimental): Oral defactinib (VS-6063) administered twice daily, in combination with intravenous paclitaxel administered on Days 1, 8, and 15 of a 28 day cycle.
  Interventions: Drug: defactinib; Drug: Paclitaxel

INTERVENTIONS:
Drug: defactinib
  Other Names: VS-6063
Drug: Paclitaxel
  Other Names: Taxol

SUMMARY:
This is a Phase I/Ib, open-label, multicenter, dose-escalation trial of paclitaxel in combination with defactinib (VS-6063), a focal adhesion kinase inhibitor, in patients with advanced ovarian cancer. This clinical study is comprised of 2 parts: Phase I (Dose Escalation) and Phase Ib (Expansion). The purpose of this study is to assess assess the safety (including the recommended phase 2 dose), the pharmacokinetics, and the anti-cancer activity of defactinib (VS-6063) when administered in combination with paclitaxel. Pharmacodynamic effects will also be examined in tumor biopsies.

ELIGIBILITY:
Inclusion Criteria:

1. Able to provide signed and dated informed consent prior to initiation of any study procedures.
2. Female subjects aged ≥ 18 years.
3. Advanced or refractory ovarian cancer, confirmed histologically.
4. Subjects may have received up to 4 prior lines of chemotherapy for their metastatic disease.
5. All persistent clinically significant toxicities from prior chemotherapy must be ≤ Grade 1.
6. ECOG performance status of 0 or 1 (refer to Appendix A), measured within 72 hours before the start of treatment.
7. Predicted life expectancy of ≥ 3 months.
8. Adequate renal function [creatinine ≤ 1.5x ULN (upper limit of normal)] or GFR of ≥ 50mL/min.
9. Adequate hepatic function (total bilirubin ≤ 1.5x ULN for the institution; AST [aspartate transaminase] and ALT [alanine transaminase] ≤ 3x ULN, or ≤ 5x ULN if due to liver involvement by tumor).
10. Adequate bone marrow function (hemoglobin ≥ 9.0 g/dL; platelets≥ 100 x109cells/L; absolute neutrophil count ≥ 1.5x109 cells/L).
11. Corrected QT interval (QTc) < 470 ms (as calculated by the Fridericia correction formula).
12. Negative pregnancy test for females of child-bearing potential; must be surgically sterile, postmenopausal, or willing and able to be compliant with a contraceptive regimen (double barrier birth control) during and for 3 months after the treatment period.
13. Willing and able to participate in the trial and comply with all trial requirements.

Exclusion Criteria:

1. Gastrointestinal (GI) condition which could interfere with the swallowing or absorption of study medication.
2. Uncontrolled or severe concurrent medical condition (including uncontrolled brain metastases). Stable brain metastases either treated or being treated with a stable dose of steroids/anticonvulsants, with no dose change within 28 days prior to the first dose of study drug, will be allowed.
3. History of upper gastrointestinal bleeding, ulceration, or perforation within 12 months prior to the first dose of study drug.
4. Known history of Gilbert's Syndrome.
5. Known history of stroke or cerebrovascular accident within 6 months prior to the first dose of study drug.
6. Subjects with known infection with human immunodeficiency virus (HIV) or Acquired Immune Deficiency Syndrome (AIDS) (testing not required).
7. Subjects with Hepatitis A, B or C (testing not required).
8. Subjects being actively treated for a secondary malignancy.
9. Cancer-directed therapy (chemotherapy, radiotherapy, hormonal therapy, biologic or immunotherapy, etc.) within 28 days of the first dose of study drug or 5 half-lives, whichever is shorter.
10. Major surgery within 28 days prior to the first dose of study drug.
11. Use of an investigational drug within 28 days or 5 half-lives (whichever is shorter) prior to the first dose of study drug. A minimum of 10 days between termination of the investigational drug and administration of the study treatment is required. In addition, any drug-related toxicity except alopecia should have recovered to grade 1 or less.
12. Pregnant or breastfeeding.
13. Any evidence of serious active infections.
14. Uncontrolled or severe cardiovascular disease, including myocardial infarct or unstable angina within 6 months prior to study treatment, New York Heart Association (NYHA) Class II or greater congestive heart failure, serious arrhythmias requiring medication for treatment, clinically significant pericardial disease, or cardiac amyloidosis.
15. Uncontrolled intercurrent illness including symptomatic congestive heart failure, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2013-02-26 (Actual); Primary Completion 2015-02-23 (Actual); Study Completion 2015-02-23 (Actual)

PRIMARY OUTCOMES:
Number of patients experiencing treatment-related adverse events as assessed by CTCAE v4.03 (Common Toxicity Criteria for Adverse Effects)during the study (safety and tolerability). | From start of treatment to end of treatment, an expected average of 12 weeks
  Adverse events and their frequency, duration and severity, as determined based on CTCAE 4.03
Determine the recommended phase 2 dose (RP2D) based on a combination of maximum tolerated dosed (MTD), review of adverse event data and review of AUC, Tmax and t1/2 obtained from PK data during the dose escalation phase of the study. | From start of treatment to end of cycle 1 (4 week cycles)
  The RP2D will be determined based on the maximum tolerated dose (MTD) of defactinib (VS-6063) in combination with paclitaxel as determined by number of participants with dose limiting toxicities (DLTs) related to defactinib in combination with paclitaxel

SECONDARY OUTCOMES:
Proportion of patients treated with paclitaxel and defactinib (VS-6063) with progression-free survival using Response Evaluation Criteria In Solid Tumors (RECIST), version 1.1 | Every 2 cycles up to end of treatment, an expected average of 12 weeks
  Response rate and progression-free survival, as determined by Response Evaluation Criteria In Solid Tumors (RECIST), version 1.1
Pharmacokinetics (PK) estimates of defactinib (VS-6063) when co-administered with paclitaxel, AUC (Area Under Curve) 0-t. | Time points at Day 1 and Day 15 in Cycle 1
  Plasma concentration of defactinib (VS-6063)
Pharmacokinetics (PK) estimates of defactinib (VS-6063) when co-administered with paclitaxel, maximum concentrations (Cmax) | Time points at Day 1 and Day 15 in Cycle 1
  Plasma concentration of defactinib (VS-6063)
Pharmacokinetics (PK) estimates of defactinib (VS-6063) when co-administered with paclitaxel, Time to maximum concentrations (Tmax) | Time points at Day 1 and Day 15 in Cycle 1
  Plasma concentration of defactinib (VS-6063)
Pharmacokinetics (PK) estimates of defactinib (VS-6063) when co-administered with paclitaxel, , estimates of concentration 1/2 life (T1/2) | Time points at Day 1 and Day 15 in Cycle 1
  Plasma concentration of defactinib (VS-6063)

OTHER OUTCOMES:
Evaluate biomarkers of defactinib (VS-6063) activity | Day 1 and Day 10 of treatment
  Pre and post dose biomarkers (including but not limited to FAK and phospho-FAK, as well as specific markers for cell cycle inhibition, apoptosis and cancer stem cells) in archival tumor tissue and new biopsy samples
Examine if the tumor expression status correlates with response to defactinib (VS-6063) therapy | From start of treatment to end of treatment, an expected average of 12 weeks
  Tumor expression status (pFAK and other biomarkers) compared with response to defactinib, as determined by Response Evaluation Criteria In Solid Tumors (RECIST), version 1.1

CONTACTS AND LOCATIONS:
Overall Officials: Hagop Youssoufian, MD, Study Chair — Verastem, Inc.
Locations (3):
- United States (3):
  - Florida Cancer Specialists, Sarasota, Florida
  - University of Oklahoma, Oklahoma City, Oklahoma
  - Sarah Cannon Research Institute, Nashville, Tennessee